CLINICAL TRIAL: NCT04078620
Title: Risk Factors for Potential Drug -Drug Interactions: Study in Surgical Intensive Care Unit -Zagazig University Hospitals
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Liza Elsayed Ali soliman shallouf, Principle investigator, Zagazig University
Other Study IDs: 4606/28-5-2018
Record Dates: First submitted 2019-08-25; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Drug Interaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Survey for drug drug interactions on medscape and lexicomp applications — Survey for drug drug interactions on Medscape and Lexicomp interaction checker applications

SUMMARY:
Drug drug interactions is frequent in critically ill patients due to polypharmacy, different drug groups and prolonged ICU or hospital stay

DETAILED DESCRIPTION:
This cross sectional study was conducted in Surgical ICU, zagazig University Hospital for 6months period.

Demographic data (age, gender),clinical history data (main diagnosis, ICU stay in days, transfer from emergency room or other departments, on mechanical ventilation or not, state of consciousness

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to Surgical ICUs for six months period

Exclusion Criteria:

* less than one day admission to ICU,not completed data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to Surgical ICUs, zagazig University Hospital
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
Severity of Drug interactions by Lexicomp interactions application | 6months period
  Lexicomp interactions classified As:
  A(no known interactions) B(no action needed) C(monitor therapy) D(consider therapy modification) X (avoid combination)
Severity of Drug interactions by Medescape interactions checker: | 6months period
  Interactions classified with Medescape interactions checker as :(contraindicated, serious use alternative, monitor closely,minor)

CONTACTS AND LOCATIONS:
Overall Officials: Liza Shallouf, Principal Investigator — Zagazig University; Heba Matar, Study Director — Zagazig University
Locations (1):
- Liza Elsayed Ali, Zagazig, Sharquia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data could be shared
Supporting Information: Study Protocol
Time Frame: For indefinite time
Access Criteria: Easy, direct information are available for other researchers